CLINICAL TRIAL: NCT02319083
Title: E-CABG: European Multicenter Study on the Outcome After Coronary Artery Bypass Grafting
Brief Title: Outcome After Coronary Artery Bypass Grafting
Acronym: E-CABG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Universita di Verona (Other); Ospedali Riuniti Trieste (Other); University of Catania (Other); University of Leicester (Other); Centre Hospitalier Universitaire de Besancon (Other); Karolinska Institutet (Other); San Camillo Hospital, Rome (Other); Rennes University Hospital (Other); S. Anna Hospital (Other); Paracelsus Medical University (Other); University of Campania Luigi Vanvitelli (Other); University of Parma (Other); University of Bari (Other); Centro Cardiologico Monzino (Other); University of Hamburg-Eppendorf (Other); University of Genova (Other)
Responsible Party: Principal Investigator, Fausto Biancari, Professor, University of Oulu
Other Study IDs: 1
Record Dates: First submitted 2014-11-23; First posted 2014-12-18 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Angina Pectoris
Keywords: CABG; Coronary artery bypass surgery; Coronary artery bypass grafting; Coronary surgery; Myocardial infarction; Coronary artery disease; Off-pump; EuroSCORE
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina Pectoris | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary artery bypass surgery: Patients undergoing coronary artery bypass surgery.
  Interventions: Procedure: Coronary artery bypass surgery

INTERVENTIONS:
Procedure: Coronary artery bypass surgery — Patients will undergo coronary artery bypass grafting
  Other Names: Coronary artery bypass grafting

SUMMARY:
The E-CABG registry is a multicenter, European registry collecting data on the preoperative characteristics, treatment strategies and outcome of patients undergoing isolated coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Improvements in the surgical treatment of coronary artery disease are possible only when implementation of current methods and development of new methods are based on the solid ground of large and reliable clinical data. Furthermore, clinical findings assume even more significance when detected in study populations from different institutions with heterogeneous referral pathways, baseline clinical characteristics and perioperative treatment strategies. The rationale of this European multicenter study is therefore to prospectively collect data on baseline characteristics, operative and anesthesiological methods and postoperative outcome of patients undergoing CABG in eleven cardiac surgery centers from five European countries. This multicenter prospective registrywill provide data to evaluate the prognostic impact of a number of patients' risk factors as well as the efficacy and safety of operative methods and drugs used during the pre-, peri- and postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of aged > 18 years undergoing isolated CABG for stable coronary artery disease or acute coronary syndrome. Patients undergoing Maze procedure will be included in this registry.

Exclusion Criteria:

* Patients undergoing any other major cardiac surgery procedure will be excluded from this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes any patient undergoing isolated coronary artery bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | The outcome measure will be assessed at time points up to 10 years after surgery
  Any death occurring after surgery

SECONDARY OUTCOMES:
Stroke | The outcome measure will be assessed at time points up to 10 years after surgery
  Any ischemic brain injury occurring after surgery and lasting > 24 hours
Prolonged use of inotropes | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of inotropes > 12 hours after surgery
Intra-aortic balloon pump | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of intra-aortic balloon pump for acute heart failure after surgery
ECMO | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of extracorporeal membrane oxygenation for acute heart failure after surgery
Repeat revascularization | The outcome measure will be assessed at time points up to 10 years after surgery
  Any repeat myocardial revascularization procedure performed after surgery
Wound infection | Participants will be followed up for 3 months after surgery
  Any deep sternal or lower limb wound infection occurring after surgery
Blood losses | Participants will be followed 12 hours after surgery
  Amont of blood losses from drainages 12 hours after surgery
Nadir hematocrit | Participants will be followed during the operation day
  Lowest hematocrit level during the operation day
Use of blood products | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Use of any blood product (red blood cell, fresh frozen plasma, Octaplas, platelets) during the in-hospital stay
Use of prothrombotic drugs | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Perioperative use of cryoprecipitate, PCC and/or rFVIIa for excessive bleeding
  PCCs
  Perioperative use of rFVIIa, PCC, cryoprecipitate
Resternotomy for bleeding | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Re-exploration for excessive bleeding
Atrial fibrillation | Participants will be followed for the duration of hospital stay (expected: 10 days)
  New episode of atrial fibrillation requiring or not cardioversion during the in-hospital stay
Renal replacement therapy | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Any renal replacement therapy during the in-hospital stay
Highest level of serum creatinine | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Highest level of serum creatinine during the in-hospital stay
Myocardial infarction | The outcome measure will be assessed at time point up to 10 years after surgery
  Myocardial infarction (diagnosed by ECG and troponin monitoring) any time after surgery
Length of stay in the intensive care unit | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Length of stay in the intensive care unit after surgery
Pericardial effusion | Participants will be followed up to 3 months after surgery.
  Pericardial effusion requiring medical or surgical treatment
Postoperative use of antibiotics | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Postoperative use of antibiotics for postoperative infection
Gastrointestinal complications | Participants will be followed for the duration of hospital stay (expected: 10 days)
  Any gastrointestinal complication requiring medical or surgical treatment after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Biancari, Professor, Study Chair — University of Oulu, Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Rubino AS, Nicolini F, Tauriainen T, Demal T, De Feo M, Onorati F, Faggian G, Bancone C, Perrotti A, Chocron S, Dalen M, Santarpino G, Fischlein T, Maselli D, Musumeci F, Santini F, Salsano A, Zanobini M, Saccocci M, Bounader K, Gatti G, Ruggieri VG, Mignosa C, Juvonen T, Mariscalco G, Biancari F. Failure to achieve a satisfactory cardiac outcome after isolated coronary surgery in low-risk patients. Interact Cardiovasc Thorac Surg. 2020 Jul 1;31(1):9-15. doi: 10.1093/icvts/ivaa062. PMID 32442254
- [Derived] Biancari F, Gatti G, Rosato S, Mariscalco G, Pappalardo A, Onorati F, Faggian G, Salsano A, Santini F, Ruggieri VG, Perrotti A, Santarpino G, Fischlein T, Saccocci M, Musumeci F, Rubino AS, De Feo M, Bancone C, Nicolini F, Kinnunen EM, Demal T, D'Errigo P, Juvonen T, Dalen M, Maselli D. Preoperative risk stratification of deep sternal wound infection after coronary surgery. Infect Control Hosp Epidemiol. 2020 Apr;41(4):444-451. doi: 10.1017/ice.2019.375. Epub 2020 Jan 20. PMID 31957634
- [Derived] Khodabandeh S, Biancari F, Kinnunen EM, Mariscalco G, Airaksinen J, Gherli R, Gatti G, Demal T, Onorati F, Faggian G, De Feo M, Santarpino G, Rubino AS, Maselli D, Salsano A, Nicolini F, Zanobini M, Ruggieri VG, Bounader K, Perrotti A, Dalen M. Perioperative Bleeding in Patients With Acute Coronary Syndrome Treated With Fondaparinux Versus Low-Molecular-Weight Heparin Before Coronary Artery Bypass Grafting. Am J Cardiol. 2019 Feb 15;123(4):565-570. doi: 10.1016/j.amjcard.2018.11.028. Epub 2018 Nov 24. PMID 30527774
- [Derived] Santarpino G, Nicolini F, De Feo M, Dalen M, Fischlein T, Perrotti A, Reichart D, Gatti G, Onorati F, Franzese I, Faggian G, Bancone C, Chocron S, Khodabandeh S, Rubino AS, Maselli D, Nardella S, Gherli R, Salsano A, Zanobini M, Saccocci M, Bounader K, Rosato S, Tauriainen T, Mariscalco G, Airaksinen J, Ruggieri VG, Biancari F. Prognostic Impact of Asymptomatic Carotid Artery Stenosis in Patients Undergoing Coronary Artery Bypass Grafting. Eur J Vasc Endovasc Surg. 2018 Nov;56(5):741-748. doi: 10.1016/j.ejvs.2018.07.042. Epub 2018 Sep 6. PMID 30197287
- [Derived] Reichart D, Rosato S, Nammas W, Onorati F, Dalen M, Castro L, Gherli R, Gatti G, Franzese I, Faggian G, De Feo M, Khodabandeh S, Santarpino G, Rubino AS, Maselli D, Nardella S, Salsano A, Nicolini F, Zanobini M, Saccocci M, Bounader K, Kinnunen EM, Tauriainen T, Airaksinen J, Seccareccia F, Mariscalco G, Ruggieri VG, Perrotti A, Biancari F. Clinical frailty scale and outcome after coronary artery bypass grafting. Eur J Cardiothorac Surg. 2018 Dec 1;54(6):1102-1109. doi: 10.1093/ejcts/ezy222. PMID 29897529
- [Derived] Mariscalco G, Rosato S, Serraino GF, Maselli D, Dalen M, Airaksinen JKE, Reichart D, Zanobini M, Onorati F, De Feo M, Gherli R, Santarpino G, Rubino AS, Gatti G, Nicolini F, Santini F, Perrotti A, Bruno VD, Ruggieri VG, Biancari F. Prior Percutaneous Coronary Intervention and Mortality in Patients Undergoing Surgical Myocardial Revascularization: Results From the E-CABG (European Multicenter Study on Coronary Artery Bypass Grafting) With a Systematic Review and Meta-Analysis. Circ Cardiovasc Interv. 2018 Feb;11(2):e005650. doi: 10.1161/CIRCINTERVENTIONS.117.005650. PMID 29440275
- [Derived] Biancari F, Brascia D, Onorati F, Reichart D, Perrotti A, Ruggieri VG, Santarpino G, Maselli D, Mariscalco G, Gherli R, Rubino AS, De Feo M, Gatti G, Santini F, Dalen M, Saccocci M, Kinnunen EM, Airaksinen JK, D'Errigo P, Rosato S, Nicolini F. Prediction of severe bleeding after coronary surgery: the WILL-BLEED Risk Score. Thromb Haemost. 2017 Feb 28;117(3):445-456. doi: 10.1160/TH16-09-0721. Epub 2016 Dec 1. PMID 27904903
- [Derived] Biancari F, Ruggieri VG, Perrotti A, Svenarud P, Dalen M, Onorati F, Faggian G, Santarpino G, Maselli D, Dominici C, Nardella S, Musumeci F, Gherli R, Mariscalco G, Masala N, Rubino AS, Mignosa C, De Feo M, Della Corte A, Bancone C, Chocron S, Gatti G, Gherli T, Kinnunen EM, Juvonen T. European Multicenter Study on Coronary Artery Bypass Grafting (E-CABG registry): Study Protocol for a Prospective Clinical Registry and Proposal of Classification of Postoperative Complications. J Cardiothorac Surg. 2015 Jun 30;10:90. doi: 10.1186/s13019-015-0292-z. PMID 26123033